CLINICAL TRIAL: NCT02915536
Title: Exploration of Effects of Excessive Iodine on Children and Tolerable Upper Intake Level of Iodine for Children
Status: Completed | Type: Observational
Sponsor: Wanqi Zhang (Other)
Collaborators: The Shandong Institute for Endemic Disease Control and Research (Unknown)
Responsible Party: Sponsor-Investigator, Wanqi Zhang, Vice Dean of School of Public Health, Tianjin Medical University, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Other Study IDs: NSFC-81273057; Nestlé Foundation (Other Grant/Funding Number: 14.03.2013); NSFC (Other Grant/Funding Number: 81273057)
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Iodine Disorders
Keywords: iodine excess; thyroid disease; children; tolerable upper intake level
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * whole blood
  * 24-h urine samples
  * spot urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Natural exposure of high iodine — Natural exposure of high iodine intake from drinking water

SUMMARY:
With the implementation of Universal Salt Iodization (USI) in 1995, China has successfully combated Iodine Deficiency Diseases (IDD). However, China is a country with a complicated iodine geographical environment with wide natural variation in the iodine content of drinking water. It has been reported that the water iodine of at least 11 provinces and cities in China is high, with nearly 31 million people exposed to the risks of excessive iodine intake. This has raised a new public health concern that a safe upper level of iodine intake should be established to ensure that people avoid ingesting excessive iodine intake while continuing to implement USI to control IDD. The investigators have successfully explored the tolerable upper intake level (UL) of iodine for Chinese adults by conducting a randomized double-blinded trial in 256 euthyroid volunteers. However, due to limited data on the safe upper intake level of iodine for children worldwide, current ULs of iodine for children are extrapolated from those for adults based on body weight or body surface area. As it is impossible to ethically conduct a randomized clinical trial regarding excessive iodine intake in children, the investigators plan an observational study to investigate children who have been living with different drinking water iodine levels for over 5 years, observing the changes of thyroid function in response to each iodine exposure level. Subtle changes in thyroid function and thyroid volume of children corresponding to different iodine intake levels will be determined, which will contribute to the establishment of UL of iodine for children.

The aim was:

1. To establish the tolerable upper intake level (UL) of iodine for children of China.
2. To define the adverse effects of excess iodine on children.
3. To monitor the iodine status of children living in high water iodine areas in China.

DETAILED DESCRIPTION:
The project is designed as a cross-sectional comparative epidemiological study, to be conducted in areas with high water iodine and adequate iodine intake, respectively. The research will include the following three stages.

First stage: In an initial contact phase of the study, workshops on the subject matter will be held in Shandong province. Regions will be sampled according to the monitoring data on water iodine collected by the Shandong Institute for Endemic Disease Control and Research, which will be a collaborative department for this study, as well as the pre-investigation. Areas in Shandong with water iodine ranging from 150μg/L to 800μg/L iodine, corresponding to urinary iodine excretion (UIE) of 300-800μg/L, will be investigated as high iodine intake areas (HI); regions with varying water iodine levels within this range will be included. Matching areas in Shandong with 10-100μg/L iodine in water, corresponding to UIE of 100-299μg/L, will be selected as the comparison areas of adequate iodine intake (AI). Refresher courses will be given to investigators and the capacity of laboratory staff will be updated. All relevant local authorities will be properly contacted. Pre-investigations will be conducted to determine the water iodine level and the former iodine status of residents, which will help the investigators to select suitable study areas. A pilot study will be conducted in a small number of subjects, including 24h urine collection and 3d dietary record to ensure that these methods are appropriate and feasible.

Second stage: A cross-sectional study of iodine intake and thyroid function in 7-14-yr-old children will be carried out. This stage mainly includes two parts.

In Part 1, 24-h and spot urinary samples (2 times) from all children will be collected to precisely evaluate the daily iodine intake of subjects. Spot urinary samples will be taken before collection of the 24-h urine samples. Teachers and parents will be trained to help children in performing the collection. 3d dietary records will be used to collect information on food and nutrient intake of participants. The parents (or guardian) and children will be trained on how to record food intake. The dietary record may be started any day of a week and correspond to the day of urine collection. The record will comprise all home food and water intake as well as out-of-home food consumption. Food frequency questionnaires (FFQ) will be used in combination with the dietary records to evaluate long-term habitual iodine intake. Simultaneously, food samples, including locally-consumed foods with relatively high iodine content and those which local residents generally consume frequently, will be sampled to determine iodine content, as will salt and water.

In Part 2, Blood samples will be collected to evaluate thyroid function and thyroid auto-antibodies, and thyroid volume of children will be detected by ultrasonography which will be conducted by professional technicians

Third stage: Iodine intake of all children will be calculated precisely and comprehensively through both 24-h UIE and dietary iodine intake (as described in Part 1). Adverse effects will be defined by parameters detected in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Native born or residents of Shandong province for at least 5 years.

Exclusion Criteria:

* Previous history of thyroid diseases or medication intake (including iodine supplements)
* protein-energy malnutrition in the long term

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: High water iodine areas in Shandong are far-ranging. An investigation in 2005 showed that water iodine content exceeded 150μg/L in 17 of the 20 counties, while water iodine in the other 3 exceeded 300μg/L. Regions with water iodine content in the range of 150-800µg/L were chosen as, with a corresponding UIE range of 300-800µg/L, were selected as high iodine intake (HI) areas for the study. Regions with water iodine content in the range of 10-100µg/L with a corresponding UIE range of 100-299µg/L were selected as adequate iodine intake (AI) study areas. Areas with high fluorine will be excluded. One to six primary schools were selected from each city by randomly sampling. Children were selected from these schools.
Sampling Method: Probability Sample
Enrollment: 2229 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
thyroid goiter confirmed by ultrasonographic thyroid volume | 1 year

SECONDARY OUTCOMES:
thyroid dysfunction confirmed by serum concentrations of FT4, FT3, and TSH with an automated chemiluminescent immunoassay by using diagnostic kits from Bayer Health Care, Siemens | 1 year

OTHER OUTCOMES:
thyroid dysfunction confirmed by serum concentrations of TPOAb and TGAb with radioimmunoassay by using kits from the Beijing North Institution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wanqi Zhang, Doctor, Study Chair — Tianjin Medical University; Jianchao Bian, Principal Investigator — The Shandong Institute for Endemic Disease Control and Research; Zuoliang Dong, Master, Principal Investigator — Tianjin Medical University; Laixiang Lin, Doctor, Principal Investigator — Tianjin Medical University; Jun Shen, Master, Principal Investigator — Tianjin Medical University; Jinbiao Wang, Principal Investigator — The Shandong Institute for Endemic Disease Control and Research; Wen Jiang, Master, Principal Investigator — The Shandong Institute for Endemic Disease Control and Research; Zhongna Sang, Doctor, Principal Investigator — Tianjin Medical University; Long Tan, Doctor, Principal Investigator — Tianjin Medical University; Wen Chen, Master, Principal Investigator — Tianjin Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teng W, Shan Z, Teng X, Guan H, Li Y, Teng D, Jin Y, Yu X, Fan C, Chong W, Yang F, Dai H, Yu Y, Li J, Chen Y, Zhao D, Shi X, Hu F, Mao J, Gu X, Yang R, Tong Y, Wang W, Gao T, Li C. Effect of iodine intake on thyroid diseases in China. N Engl J Med. 2006 Jun 29;354(26):2783-93. doi: 10.1056/NEJMoa054022. PMID 16807415
- [Background] Laurberg P, Bulow Pedersen I, Knudsen N, Ovesen L, Andersen S. Environmental iodine intake affects the type of nonmalignant thyroid disease. Thyroid. 2001 May;11(5):457-69. doi: 10.1089/105072501300176417. PMID 11396704
- [Background] Izzeldin HS, Crawford MA, Jooste PL. Population living in the Red Sea State of Sudan may need urgent intervention to correct the excess dietary iodine intake. Nutr Health. 2007;18(4):333-41. doi: 10.1177/026010600701800403. PMID 18087865
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Laurberg P, Pedersen KM, Hreidarsson A, Sigfusson N, Iversen E, Knudsen PR. Iodine intake and the pattern of thyroid disorders: a comparative epidemiological study of thyroid abnormalities in the elderly in Iceland and in Jutland, Denmark. J Clin Endocrinol Metab. 1998 Mar;83(3):765-9. doi: 10.1210/jcem.83.3.4624. PMID 9506723
- [Background] Laurberg P, Cerqueira C, Ovesen L, Rasmussen LB, Perrild H, Andersen S, Pedersen IB, Carle A. Iodine intake as a determinant of thyroid disorders in populations. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):13-27. doi: 10.1016/j.beem.2009.08.013. PMID 20172467
- [Background] Su X., Liu S., Shen H., Zhang S., Wei H., Yu J., Ye Y., Li Y., Liu Y., Zhang Z., Sun D. National iodine deficiency disorder surveillance: a sum up of data in 2005 and an analysis. Chinese Journal of Endemiology. 2007, 26(1): 67-69.
- [Background] Zimmermann MB, Andersson M. Assessment of iodine nutrition in populations: past, present, and future. Nutr Rev. 2012 Oct;70(10):553-70. doi: 10.1111/j.1753-4887.2012.00528.x. PMID 23035804
- [Background] Pearce EN, Gerber AR, Gootnick DB, Khan LK, Li R, Pino S, Braverman LE. Effects of chronic iodine excess in a cohort of long-term American workers in West Africa. J Clin Endocrinol Metab. 2002 Dec;87(12):5499-502. doi: 10.1210/jc.2002-020692. PMID 12466344
- [Background] Burgi H. Iodine excess. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):107-15. doi: 10.1016/j.beem.2009.08.010. PMID 20172475
- [Background] Zimmermann MB, Ito Y, Hess SY, Fujieda K, Molinari L. High thyroid volume in children with excess dietary iodine intakes. Am J Clin Nutr. 2005 Apr;81(4):840-4. doi: 10.1093/ajcn/81.4.840. PMID 15817861
- [Background] Ergur AT, Evliyaoglu O, Siklar Z, Bilir P, Ocal G, Berberoglu M. Evaluation of thyroid functions with respect to iodine status and TRH test in chronic autoimmune thyroiditis. J Clin Res Pediatr Endocrinol. 2011;3(1):18-21. doi: 10.4274/jcrpe.v3i1.04. Epub 2011 Feb 23. PMID 21448329
- [Background] Shen H., Zhang S., Liu S., Su X., Shen Y., Han H. Study on the geographic distribution of national high water iodine areas and the contours of water iodine in high iodine areas. Chinese Journal of Endemiology. 2007, 26(6): 658-661.
- [Background] Guo X., Wang X., Liu Y., Huang J., Zhai L., Chen Z. Investigation of distribution of high water iodine areas of northwestern Shandong and the current status of inhabitant edible salt. Chinese Journal of Preventive Medicine. 2005, 39(2): 77-78.
- [Background] WHO/UNICEF/ICCIDD. Assessment of iodine deficiency disorders and monitoring their elimination. 3rd ed. Geneva, 2007.
- [Background] Lv S, Zhao J, Xu D, Chong Z, Jia L, Du Y, Ma J, Rutherford S. An epidemiological survey of children's iodine nutrition and goitre status in regions with mildly excessive iodine in drinking water in Hebei Province, China. Public Health Nutr. 2012 Jul;15(7):1168-73. doi: 10.1017/S1368980012000146. Epub 2012 Feb 8. Erratum In: Public Health Nutr. 2014 Nov;17(11):2624. Chong, Zhengshui [corrected to Chong, Zhenshui]. PMID 22314228
- [Background] National Health and Medical Research Council. Nutrient reference values for Australia and New Zealand including recommended dietary intakes. 2005.
- [Background] Chen W, Sang ZN, Liu H, Shen J, Zhao N, Tan L, Wei W, Zhang GQ, Wen SC, Zhang WQ. [Investigation of thyroid function abnormalities in children in high water iodine areas of Hebei province]. Zhonghua Yu Fang Yi Xue Za Zhi. 2012 Feb;46(2):148-51. Chinese. PMID 22490198
- [Background] Shen H, Liu S, Sun D, Zhang S, Su X, Shen Y, Han H. Geographical distribution of drinking-water with high iodine level and association between high iodine level in drinking-water and goitre: a Chinese national investigation. Br J Nutr. 2011 Jul;106(2):243-7. doi: 10.1017/S0007114511000055. PMID 21320367
- [Result] Chen W, Wu Y, Lin L, Tan L, Shen J, Pearce EN, Guo X, Wang W, Bian J, Jiang W, Zhang W. 24-Hour Urine Samples Are More Reproducible Than Spot Urine Samples for Evaluation of Iodine Status in School-Age Children. J Nutr. 2016 Jan;146(1):142-6. doi: 10.3945/jn.115.215806. Epub 2015 Nov 25. PMID 26609173
- [Derived] Cui T, Wang W, Chen W, Pan Z, Gao S, Tan L, Pearce EN, Zimmermann MB, Shen J, Zhang W. Serum Iodine Is Correlated with Iodine Intake and Thyroid Function in School-Age Children from a Sufficient-to-Excessive Iodine Intake Area. J Nutr. 2019 Jun 1;149(6):1012-1018. doi: 10.1093/jn/nxy325. PMID 31070733
- [Derived] Chen W, Zhang Q, Wu Y, Wang W, Wang X, Pearce EN, Tan L, Shen J, Zhang W. Shift of Reference Values for Thyroid Volume by Ultrasound in 8- to 13-Year-Olds with Sufficient Iodine Intake in China. Thyroid. 2019 Mar;29(3):405-411. doi: 10.1089/thy.2018.0412. PMID 30696370
- [Derived] Chen W, Zhang Y, Hao Y, Wang W, Tan L, Bian J, Pearce EN, Zimmermann MB, Shen J, Zhang W. Adverse effects on thyroid of Chinese children exposed to long-term iodine excess: optimal and safe Tolerable Upper Intake Levels of iodine for 7- to 14-y-old children. Am J Clin Nutr. 2018 May 1;107(5):780-788. doi: 10.1093/ajcn/nqy011. PMID 29722836
- [Derived] Chen W, Li X, Wu Y, Bian J, Shen J, Jiang W, Tan L, Wang X, Wang W, Pearce EN, Zimmermann MB, Carriquiry AL, Zhang W. Associations between iodine intake, thyroid volume, and goiter rate in school-aged Chinese children from areas with high iodine drinking water concentrations. Am J Clin Nutr. 2017 Jan;105(1):228-233. doi: 10.3945/ajcn.116.139725. Epub 2016 Dec 7. PMID 27927635